CLINICAL TRIAL: NCT02251431
Title: MB001-067 A PROSPECTIVE, DOUBLE BLIND, PLACEBO CONTROLLED, PARALLEL GROUP, RANDOMIZED TRIAL OF EXTENDED RELEASE EXENATIDE VERSUS PLACEBO (COHORT A) AND A PROSPECTIVE, SINGLE GROUP, OPEN-LABEL, BLINDED OUTCOME TRIAL OF EXTENDED RELEASE EXENATIDE (COHORT B) IN DIABETIC PATIENTS WITH TYPE 4 CARDIORENAL SYNDROME (EXTEND-CRS TRIAL) AMENDMENT 3
Brief Title: Extended Release Exenatide Versus Placebo In Diabetic Patients With Type 4 Cardiorenal Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 014-149; D5551L00004/ISSEXEN0013 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2014-09-12; First posted 2014-09-29 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease; Left Ventricular Diastolic Dysfunction
Keywords: diabetes mellitus; chronic kidney disease; diastolic function; cardiac fibrosis; cardiac strain; cardiac biomarker; renal biomarker
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Ventricular Dysfunction, Left; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide-extended release (Experimental): Exenatide-extended release (BYDUREON™) 2 mg subcutaneously once per week x 38 weeks
  Interventions: Drug: BYDUREON
- Placebo (Placebo Comparator): Matching placebo subcutaneously once per week x 38 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BYDUREON — Exenatide-extended release, Cohorts A and B
  Arms: Exenatide-extended release
Drug: Placebo — Cohort A only
  Other Names: Matching placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
Among adult individuals with type 2 diabetes mellitus and at risk for heart failure with impaired relaxation of the heart mildly reduced kidney filtration function (Type 4 cardiorenal syndrome) this trial will evaluate the quantitative impact of 38 weeks of treatment with exenatide extended-release injections versus placebo. on a cardiac biomarker blood test score, cardiac fibrosis seen on magnetic resonance scanning, cardiac strain identified by ultrasonography and strain rate imaging, and a kidney urine biomarker score.

DETAILED DESCRIPTION:
Primary Aim

Among adult individuals with type 2 diabetes mellitus (T2DM) and at risk for diastolic heart failure (DHF) and mildly reduced renal filtration function (Type 4 cardiorenal syndrome), to evaluate the quantitative impact on the MISS (myocardial injury summary score) cardiac biomarker score, cardiac fibrosis by MRI, cardiac strain by ultrasonography and strain rate imaging, and KISS (kidney injury summary score) kidney biomarker score after 38 weeks of treatment with exenatide extended-release or placebo.

Secondary Aim

To evaluate the inter-relationships between demographic, clinical, and biochemical variables (MISS score, KISS score) and of progressive cardiac fibrosis as assessed by MRI, strain-rate imaging, and in adult individuals with T2DM and at risk for DHF (Type 4 cardiorenal syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Type 2 diabetes mellitus with hemoglobin A1C 6.6-9.9% with or without the use of insulin
* Estimated glomerular filtration rate (eGFR) between 50 and 90 ml/min/1.73 m2

Exclusion Criteria:

* Allergy or intolerance to gadolinium
* Implanted cardiac pacemaker, defibrillator, loop recorder, or other implanted metallic device
* Any other metallic implanted device that is a contra-indication to MRI scanning
* eGFR < 50 ml/min/1.73 m2
* eGFR > 90 ml/min/1.73 m2
* Patient has ever been treated with an approved or investigational GLP-1 receptor agonist e.g. BYETTA™ (exenatide), BYDUREON™ (Exenatide extended-release), VICTOZA™ (liraglutide), or taspoglutide
* Patient is enrolled in another experimental protocol which involves the use of an investigational drug or device, or an intervention that would interfere with the conduct of the trial.
* Disorders of iron metabolism
* Collagen vascular diseases
* Myocardial infarction
* Use of DDP4 inhibitors, and PPAR gamma agonists
* Pregnancy or planned pregnancy during the trial period
* Hemoglobin A1C of ≥ 10.0% or <6.6%
* Fasting glucose ≥ 260 mg/dl
* Clinically significant abnormal baseline laboratories
* Morbid obesity or body girth that prohibits the ability to undergo echocardiography or MRI scanning with high-quality image results
* Renal transplantation
* Severe gastrointestinal, liver, or neurodegenerative disease
* Decompensated liver cirrhosis (Child-Pugh score >7)
* New York Heart Association Class III or IV heart failure
* Patients have alanine aminotransaminase (ALT) greater than 5 times the upper limit of the reference range.
* Prior pancreatitis
* Personal or family history of medullary thyroid adenoma or carcinoma (MTC)
* Multiple Endocrine Neoplasia syndrome type 2 (MEN 2).
* History of severe hypoglycemia
* Prior bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A McCullough, MD, MPH, Study Chair — Baylor Research Institute
Locations (1):
- Baylor Scott and White Research Institute- Baylor Heart and Vascular Hospital, Dallas, Texas, United States

REFERENCES:
- [Background] Chinnaiyan KM, Alexander D, Maddens M, McCullough PA. Curriculum in cardiology: integrated diagnosis and management of diastolic heart failure. Am Heart J. 2007 Feb;153(2):189-200. doi: 10.1016/j.ahj.2006.10.022. PMID 17239676
- [Background] Davidson MH. Cardiovascular effects of glucagonlike peptide-1 agonists. Am J Cardiol. 2011 Aug 2;108(3 Suppl):33B-41B. doi: 10.1016/j.amjcard.2011.03.046. PMID 21802579
- [Background] Levine GD, Rosai J, Bearman RM, Polliack A. The fine structure of thymoma, with emphasis on its differential diagnosis. A study of ten cases. Am J Pathol. 1975 Oct;81(1):49-86. PMID 1080957
- [Background] Best JH, Hoogwerf BJ, Herman WH, Pelletier EM, Smith DB, Wenten M, Hussein MA. Risk of cardiovascular disease events in patients with type 2 diabetes prescribed the glucagon-like peptide 1 (GLP-1) receptor agonist exenatide twice daily or other glucose-lowering therapies: a retrospective analysis of the LifeLink database. Diabetes Care. 2011 Jan;34(1):90-5. doi: 10.2337/dc10-1393. Epub 2010 Oct 7. PMID 20929995
- [Background] McCullough PA, Olobatoke A, Vanhecke TE. Galectin-3: a novel blood test for the evaluation and management of patients with heart failure. Rev Cardiovasc Med. 2011;12(4):200-10. doi: 10.3909/ricm0624. PMID 22249510
- [Background] Wang YC, Yu CC, Chiu FC, Tsai CT, Lai LP, Hwang JJ, Lin JL. Soluble ST2 as a biomarker for detecting stable heart failure with a normal ejection fraction in hypertensive patients. J Card Fail. 2013 Mar;19(3):163-8. doi: 10.1016/j.cardfail.2013.01.010. PMID 23482076
- [Background] Jellis C, Martin J, Narula J, Marwick TH. Assessment of nonischemic myocardial fibrosis. J Am Coll Cardiol. 2010 Jul 6;56(2):89-97. doi: 10.1016/j.jacc.2010.02.047. PMID 20620723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide-extended Release | Placebo
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 57 patients were enrolled from November 2015 to December 2019. Despite original plan of enrolling 104 patients, the recruitment stopped early due to poor accrual
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide-extended Release | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.78 (12.83) | 55.17 (9.64) | 56.50 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Diabetes [Count of Participants; unit: Participants] | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Galectin-3
Description: Mean change in plasma galectin-3 (pg/ml)
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
pg/ml
  Baseline | 9570.91 (4990.06) | 9266.7 (6032.8)
  End of study (38th week) | 9539.21 (3893.04) | 8098.78 (6272.55)

2. Primary Outcome: ST2
Description: Mean change in plasma ST2 (pg/ml)
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
pg/ml
  Baseline | 635.2 (449.82) | 443.18 (380.34)
  End of study (38th week) | 524.68 (423.61) | 534.53 (302.89)

3. Primary Outcome: NGAL
Description: Mean change in urine neutrophil gelatinase associated lipocalin (NGAL):creatinine (Cr) ratio
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 17.35 (29.01) | 18.44 (25.01)
  End of study (38th week) | 14.01 (14.87) | 24.39 (40.37)

4. Primary Outcome: KIM-1
Description: Mean change in urine kidney injury molecule-1 (KIM-1):Cr ratio
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 0.1 (0.08) | 0.13 (0.09)
  End of study (38th week) | 0.13 (0.14) | 0.1 (0.05)

5. Primary Outcome: L-FABP
Description: Mean change in urine L-type fatty acid binding protein:Cr ratio
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 2.61 (3.72) | 3.24 (4.17)
  End of study (38th week) | 2.05 (2.18) | 3 (2.85)

6. Primary Outcome: IL-18
Description: Mean change in urine interleukin-18:Cr ratio
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: pg/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
pg/mmol Creat
  Baseline | 1.68 (2.4) | 3.48 (4.69)
  End of study (38th week) | 1.96 (3.5) | 2.68 (2.48)

7. Primary Outcome: Alpha GST
Description: Mean change in urine alpha glutathione S-transferase (αGST):Cr ratio
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 0.06 (0.2) | 0.67 (1.83)
  End of study (38th week) | 0.05 (0.16) | 0.27 (0.56)

8. Primary Outcome: Troponin I
Description: Mean change in plasma ultrasensitive troponin I (pg/ml)
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
pg/ml
  Baseline | 230.85 (282.73) | 415.65 (446.33)
  End of study (38th week) | 238.53 (283.59) | 504.48 (599.4)

9. Primary Outcome: Pi GST
Description: Mean change in pi glutathione S-transferase (piGST):Cr ratio
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 2.2 (3.41) | 3.99 (3.96)
  End of study (38th week) | 3.03 (5.67) | 4.27 (4.67)

10. Primary Outcome: NAG
Description: Mean change in urine N-acetyl-β-D-glucosaminidase (NAG):Cr ratio
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 17.35 (29.01) | 18.44 (25.01)
  End of study (38th week) | 14.01 (14.87) | 24.39 (40.37)

11. Primary Outcome: Cystatin-C
Description: Mean paired change in urine cystatin-C:Cr ratio (uCysC:Cr)
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 2.07 (2.64) | 1.84 (1.19)
  End of study (38th week) | 1.47 (1.22) | 1.57 (1.17)

12. Primary Outcome: BNP
Description: Mean change in plasma B-type natriuretic peptide BNP (pg/ml)
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
pg/ml
  Baseline | 4.87 (9.3) | 9.88 (14.52)
  End of study (38th week) | 5.59 (9.59) | 14.02 (22.53)

13. Primary Outcome: ACR
Description: Mean change in urine albumin:Cr ratio (ACR)
Time Frame: 38 weeks
Measure: Mean (Standard Deviation); unit: ng/mmol Creat
Arm/Group | Exenatide-extended Release | Placebo
Number analyzed (Participants) | 29 | 28
ng/mmol Creat
  Baseline | 6678.23 (12662.79) | 9713.65 (14380.38)
  End of study (38th week) | 3963.49 (3101.13) | 9825.2 (9539.34)

ADVERSE EVENTS:
Time Frame: 38 weeks from study initiation
Arm/Group | Exenatide-extended Release | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/28
Other Adverse Events (participants affected / at risk) | 20/29 | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide-extended Release (N=29) | Placebo (N=28)
NSTEMI (non ST elevated myocardial infarction) (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide-extended Release (N=29) | Placebo (N=28)
Injection site reaction (General disorders) | 15 (28) | 10 (13)
Gastrointestinal events, myalgia, fatigue (Gastrointestinal disorders) | 20 (61) | 21 (107)

LIMITATIONS AND CAVEATS:
Our recruitment stopped early due to low accrual rate. Hence, null findings may be a result of lack of statistical power. Accordingly, our results should be interpreted as hypothesis-generating.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT02251431/Prot_SAP_000.pdf